CLINICAL TRIAL: NCT04144387
Title: Evaluation of the Impact of the Update Multiple Myeloma Criteria on the Natural History of Smoldering Myeloma in Order to Establish New Recommendations About Follow-up and Prognostic Evaluation of Smoldering Myeloma (CARRISMM)
Brief Title: Evaluation of the Impact of the Update SMM Criteria on the Natural History of SMM to Establish New Recommendations.
Acronym: CARRISMM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IFM 2017-04; 2016-002650-20 (Other: IDRCB Number)
Record Dates: First submitted 2019-10-18; First posted 2019-10-30 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — Myelography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): Each patient included in the study will be followed for 5 years
  Interventions: Procedure: Myelogram

INTERVENTIONS:
Procedure: Myelogram — Two additional myelograms will be performed comparing to standard of care.

SUMMARY:
This study is a prospective open label interventional multicenter study evaluating the impact of the update multiple myeloma criteria on the natural history of smoldering myeloma in order to establish new recommendations about follow up and prognostic evaluation of smoldering myeloma.

DETAILED DESCRIPTION:
In 2014, the International Myeloma Working Group (IMWG) proposed a revised classification of multiple myeloma (MM) and smoldering myeloma (SMM). Since the new definition of SMM proposed excludes "ultra-high risk SMM", the evolution profile of SMM will change. Therefore, investigators need to update their knowledge of SMM to optimize the management of patients. This project is expected to describe more precisely the new landscape of SMM.

The results will help to establish new recommendations for the standard care of SMM and especially for defining accurate follow-up and risk stratifying.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* SMM defined by IMWG 2014 criteria

  1. Serum monoclonal protein (IgG or IgA) ≥30 g/L and/or urinary monoclonal protein ≥500 mg per 24 h and/or clonal bone marrow plasma cells 10-60%
  2. Absence of myeloma defining events or amyloidosis
* Diagnosed less than 1 year before the inclusion
* Able and willing to give valid written informed consent. Patients must give written informed consent (IC) in accordance with institutional and local guidelines.

Exclusion Criteria:

* Previous antimyeloma treatment including bisphosphonates
* Second Primary Malignancy and/or auto-immune disease treated by immunosuppressive drugs.
* Evidence of end organ damage that can be attributed to the underlying SMM:

  1. Hypercalcaemia: serum calcium >0.25 mmol/L (>10 mg/L) higher than the upper limit of normal or >2.75 mmol/L (>110 mg/L)
  2. Renal insufficiency: creatinine clearance <40 mL/min or serum creatinine >177 μmol/L (>20 mg/L)
  3. Anaemia: haemoglobin value of >2 g/dL below the lower limit of normal, or a haemoglobin value <10 g/dL
  4. Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or Positron Emission Tomography-Computed Tomography (PET-CT)
* Presence of one of the following biomarkers of malignancy:

  1. Clonal bone marrow plasmocytosis ≥60%
  2. Involved/uninvolved serum Free Light Chain (FLC) ratio ≥ 100 (The involved free light chain must be ≥100 mg/L)
  3. Presence of one or more focal lesions on MRI studies (each focal lesion must be 5 mm or more in size)
* History of malignancy other than SMM within 3 years before inclusion
* Amyloidosis
* POEMS syndrome
* Contraindication to MRI
* Pregnancy
* Nursing mother
* Legally protected adults (under judicial protection, guardianship, or supervision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Assess the annual risk estimated at 2 years of progression from SMM to MM | 2 years
  Progression to MM will be defined, according to IMWG 2014 revised classification, by the apparition of one or more myeloma defining events:
  * Evidence of end organ damage that can be attributed to the underlying MM (CRAB criteria)
  * Presence of one of the following biomarkers of malignancy (new criteria of MM introduced in 2014 IMWG recommendations)

SECONDARY OUTCOMES:
Assess the risk of progression to MM evaluating biological factors | 5 years
  * Progression of monoclonal component level (serum M component, urine M component or FLC involved/uninvolved) defined by increase of ≥ 25% from inclusion value.
  * Progression of percentage of phenotypically abnormal Bone Marrow Plasma Cells defined by increase of ≥ 10 % from inclusion value or an increase to over 95%
Assess the risk of progression to MM evaluating radiological markers | 5 years
  MRI progression : Progression of MRI abnormalities defined by any one or more of the following
  * Appearance of new focal lesion or new diffuse infiltration of previously unaffected regions
  * Growth of previously preexisting < 5mm focal(s) lesion(s)
  * Progressive diffuse infiltration of already affected bones
Describe the clonal and sub-clonal evolution of SMM | 5 years
  Genetic analysis of bone marrow plasma cells at inclusion and during follow up to give data about the clonal and subclonal evolution of SMM (analysis of the mutations present in the tumor plasma cells, the allele frequency of each mutations, the determination of the clonal evolution mode for patients who will evolve to overt MM, the evaluation of copy number changes enabling to detect all the prognostic changes (1p32, 1q, 17p13), and (v) all the 14q32 translocations).
Describe annual risk of progression from SMM to MM at 5 years | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Olivier Decaux, Principal Investigator — Rennes University Hospital
Locations (90):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Institut Jules Bordet, Brussels
  - CHU UCL Namur ASBL Site Godinne, Yvoir
- France (86):
  - Centre Hospitalier, Abbeville
  - CHU Amiens Sud, Amiens
  - CHRU - Hôpital du Bocage, Angers
  - Ch Annecy Genevois, Annecy
  - Centre Hospitalier d'Argenteuil Victor Dupouy, Argenteuil
  - CH d'Arras, Arras
  - Centre Hospitalier de Auch, Auch
  - Centre Hospitalier H. Duffaut, Avignon
  - Centre hospitalier de la Côte Basque, Bayonne
  - Hôpital Nord Franche Comté, Belfort
  - Centre Hospitalier Simone Veil, Blois
  - Hôpital Avicenne, Bobigny
  - Institut Bergonié - Pavillon Saint Genès - 1er étage, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre hospitalier Pierre Oudot, Bourgoin
  - CHRU Brest - Hôpital A. Morvan, Brest
  - CHU Caen - Côte de Nacre, Caen
  - Centre Hospitalier, Cannes
  - CH René Dubos, Cergy-Pontoise
  - Médipôle de Savoie, Challes-les-Eaux
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - CH Chambéry, Chambéry
  - Hôpital d'Instruction des Armées Percy, Clamart
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - Centre Hospitalier, Dax
  - CHU François Mitterand, Dijon
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Hôpital de Fréjus, Fréjus
  - CHU de Grenoble, Grenoble
  - Institut Daniel Hollard, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Groupe Hospitalier de La Rochelle, La Rochelle
  - Hospital Jacques Monod, Le Havre
  - Centre Hospitalier, Le Mans
  - Centre Hospitalier, Lens
  - Centre hospitalier Robert Boulin, Libourne
  - CHRU Hôpital Claude Huriez, Lille
  - Centre Hospitalier Universitaire (CHU) de Limoges, Limoges
  - Hôpital du Scorff, Lorient
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Léon Bérard, Lyon
  - CH Meaux, Meaux
  - Hospital Sainte Blandine, Metz
  - Hôpital de Mercy (CHR Metz-Thionville), Metz
  - Centre de Recherche Clinique / GHT des Landes, Mont-de-Marsan
  - Clinique du Parc, Montpellier
  - Hopital Saint Eloi - CHU Montpellier, Montpellier
  - Hôpital E. Muller, Mulhouse
  - CHRU Hôpitaux de Brabois, Nancy
  - Centre Catherine de Sienne, Nantes
  - CHRU Hôtel Dieu, Nantes
  - Hôpital Archet 1, Nice
  - CHU Carémeau, Institut de Cancérologie du Guard, Nîmes
  - CH La Source, Orléans
  - CHU Hôpital Saint Antoine, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - Hôpital Saint Louis, Paris
  - La Pitié, Paris
  - CH Saint Jean, Perpignan
  - CHRU - Hôpital du Haut Lévêque - Centre François Magendie, Pessac
  - Centre Hospitalier de Perigueux, Périgueux
  - CHU Poitiers - Pôle régional de Cancérologie, Poitiers
  - Centre Hospitalier de Quimper Cornouaille, Quimper
  - Hôpital Robert Debré, Reims
  - CHRU Hôpital de Pontchaillou, Rennes
  - Hôpital Privé Sévigné, Rennes
  - Centre Hospitalier Jacques Puel, Rodez
  - CH Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest
  - Centre Hospitalier, Saint-Quentin
  - CH Saint Malo, St-Malo
  - CHU Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Strasbourg Oncologie Libérale, Strasbourg
  - Centre hospitalier de Tarbes, Tarbes
  - Hôpital Inter-Armées Ste Anne, Toulon
  - Pôle IUCT Oncopole CHU, Toulouse
  - CHRU Hôpital Bretonneau - Centre Henry Kaplan, Tours
  - Centre Hospitalier de Troyes, Troyes
  - Centre Hospitalier de Valence, Valence
  - Centre Hospitalier, Valenciennes
  - CH Bretagne Atlantique Vannes et Auray - P. Chubert, Vannes
  - CHV André Mignot - Université de Versailles, Versailles
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No